CLINICAL TRIAL: NCT01972386
Title: Spectrum Image Analysis of Lymph Nodes During Endobronchial Ultrasound-Guided (EBUS) Transbronchial Needle Aspiration (TBNA) in Patients With Lung Cancer
Brief Title: EBUS/Spectrum Analysis
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 12-5898-CE
Record Dates: First submitted 2013-10-08; First posted 2013-10-30 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Spectrum Image Analysis
  Interventions: Device: Spectrum Image Analysis using a Linear Array Ultrasound Bronchoscope

INTERVENTIONS:
Device: Spectrum Image Analysis using a Linear Array Ultrasound Bronchoscope

SUMMARY:
To evaluate the clinical benefit of spectrum analysis of endobronchial ultrasound images of lymph nodes during EBUS TBNA for lymph node staging in patients with lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 years or older
* Patients with known or suspected lung cancer who require EBUS-TBNA for lymph node staging

Exclusion Criteria:

* Patients who are deemed on clinical grounds not to be medically fit for a bronchoscopy
* Inability to give informed consent
* Patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lung cancer or suspected lung cancer who undergo EBUS TBNA for lymph node staging.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2013-09; Primary Completion 2015-09 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Lymph Node Staging | Pathology report will be completed as soon as possible after the procedure. (Within one year)
  The lymph node staging will be determined by the pathology report of the biopsy taken from the patients lymph node(s).

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada